Efficacy of the Transition of the Foot Strike Pattern From Rearfoot to Midfoot or Forefoot During Running on Pain and Disability in Cadets With Chronic Musculoskeletal Pain

NCT ID not yet assingned

## 06/11/2019

## **Informed Consent Form**

You are being invited to participate in the research "Efficacy of the transition from the rearfoot pattern to the forefoot or midfoot during the race in reducing pain and disability in cadets of Naval School with chronic musculoskeletal pain: a randomized controlled trial."

Your participation is not mandatory. At any time you may withdraw your participating and withdraw your consent. Your refusal will not cause any damage to your relationship with the Naval Researcher or School and no penalty.

The objectives of this study are to compare the efficacy of altering the pattern of how the foot strike pattern the ground during the run with the muscular strengthening performances in cadets Naval School with musculoskeletal pain in the lumbar and lower limbs associated with running.

Your participation in this research will consist of data that will be used from the questionnaires you fill out with data on location of pain, duration, frequency, and shooting of the running in order to evaluate the way you run. This footage will be performed by the military of the Physiotherapy sector of this place and will be accessible only by the researchers. After filming, if you have the criteria for inclusion in the study, you will be randomly included in one of three groups. All groups will be offered the standard treatment of the physiotherapy sector. This treatment includes techniques of thermotherapy, laser therapy and electrotherapy. One group will receive only standard care from the physiotherapy sector. The second group will perform specific muscular strengthening exercises for musculoskeletal pain in the lumbar spine and lower limbs. The third group will perform the change of the foot strike pattern on the ground during the race. The interventions of all groups will be carried out under the guidance of the physiotherapist researcher at the Naval School. The allocation of the participant in the group is random and the researcher has no influence on the designation of the participants in the groups. If one therapeutic approach is superior to the other, the research physiotherapist undertakes to offer the most effective treatment to the participants who were allocated to another group after the research was completed.

Filming, standard physiotherapeutic treatment, muscle strengthening exercises and the transition of the tread will be performed within the period reserved for the practice of physical exercises, not impairing their curriculum. Participants will not have any research-related expenses. The data collected will be used only for medical evaluation parameters and will not be used for any academic evaluation of the Naval School.

The risks they will be exposed to are: worsening of musculoskeletal pain and risk of falls at the moment of the run during the transition from the foot to the forefoot, in addition to the risks to which they are already exposed during the physical activity they routinely practice. Nurses, doctors and ambulances will be made available throughout their participation in the research in order to assist in the aforementioned risks.

The benefits related to your participation are:

- Analysis of the race movement to identify possible changes in movement that may be the origin of musculoskeletal pain;
- Possibility of improvement of musculoskeletal pain through the therapeutic approach of any of the groups.

The participant will be entitled to full indemnity in case of any damage related to the research during or after the realization of the same, in accordance with Resolution 466/2012 of the National Health Council.

The information obtained through this research will be confidential and we will ensure the confidentiality of your participation. The data will not be disclosed in order to enable its identification. You will receive a copy of this term, where the phone number and the principal address of the principal researcher and CEP can be found, and you can ask questions about the project and its participation, now or at any time.

Thais de Freitas Borba Pinheiro

Avenida Almirante Silvio de Noronha s / n Castelo - Rio de Janeiro, RJ CEP 20021-010.

Phones (21) 3974-1548 / (21) 99806-0266

I declare that I have understood the objectives, risks and benefits of my participation in the research and agree to participate.

I authorize the use of my photo or filming in the research for presentation in thesis, congress or publication in a scientific journal in which it will not be possible to identify the participant.

Name and signature of research volunteer